CLINICAL TRIAL: NCT06205537
Title: Effects of Nutritional Ingredients on Muscle Health and Recovery Following a Short Bout of Exhaustive Exercise in Older Adults
Brief Title: Muscle Health and Recovery in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BL78
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Exercise Induced Muscle Damage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Liquid Supplement (ONS) Group A (Placebo Comparator): One 8 oz. serving
  Interventions: Other: Control Liquid Supplement
- Oral Liquid Supplement (ONS) Group B (Experimental): One 8 oz. serving
  Interventions: Other: Experimental Liquid Supplement

INTERVENTIONS:
Other: Control Liquid Supplement — Ready to drink supplement.
  Arms: Oral Liquid Supplement (ONS) Group A
Other: Experimental Liquid Supplement — Ready to drink supplement.
  Arms: Oral Liquid Supplement (ONS) Group B

SUMMARY:
This is a prospective, randomized, placebo controlled, double-blinded study to evaluate the efficacy of a combination of nutritional ingredients on muscle health and recovery from a short bout of exhaustive exercise in healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant, male and female (≥60 and ≤75 years of age)
* Subject is ambulatory
* Body mass index (BMI) >18.5 but <30 kg/m2
* Subject agrees to refrain from starting an exercise program throughout the trial
* Has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), and applicable privacy regulation authorization prior to any participation in the study
* Willingness to follow the protocol as described, including consumption of study product per the protocol, and completing any forms/questionnaires needed throughout the study

Exclusion Criteria:

* Subject reports having type 1 or type 2 diabetes
* Subject reports having undergone major surgery that might affect the outcomes
* Has stated presence of partial or full lower artificial limb
* Is unable to participate in an exercise protocol
* Habitually engages in strenuous exercise, duration of 1 hour or longer, 3 or more times per week
* Subjects has received systemic corticosteroid treatment in the last 3 months
* Subject reports recent oral antibiotic use
* Subject reports of current active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix
* Subject reports of significant cardiovascular event within 6 months prior to study entry or history of congestive heart failure
* Subject reports of end-stage organ failure or is post-organ transplant
* Subject reports of current or history of renal disease or severe gastroparesis
* Subject reports of current diagnosed hepatic disease
* Subject reports of history of GI disease that could impact digestion or absorption of the study product
* Subject reports a history of autoimmune or connective tissue diseases that may affect muscle.
* Subject reports clotting or bleeding disorders.
* Subject reports a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis A, B or C, or HIV.
* Subjects reports an eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Subject reports having statin-induced myopathy at time of screening.
* Subject reports taking certain dietary supplements, oral nutritional supplements or high protein nutritional supplements, or medications, that could profoundly affect muscle metabolism. Exceptions for multi-vitamin/mineral supplement and inhaled steroids for asthma, topical or optical steroids. Those users who can stop using such products for ≥4 weeks before baseline visit and agree to refrain from taking them over the study period need not be excluded.
* Subject cannot refrain from using specific oils in their home cooked meals over the course of the study.
* Has an allergy or intolerance to any ingredient in the study product.
* Participates in another study that has not been approved as a concomitant study by Abbott Nutrition.
* Subject has participated in another research study in the last 3 months that involved an inconvenience allowance or biosampling (including >50ml blood or any tissue samples).

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Leg Strength | Pre-Exercise (Day -1) to Post Exercise Recovery (up to 7 Days)
  Change in Peak torque of maximum voluntary contraction (MVC)

SECONDARY OUTCOMES:
Muscle Fatigue | Pre-Exercise (Day -1) to Post Exercise Recovery (up to 7 Days)
  Time to failure during a sub-maximal isometric contraction of the knee extensors
Muscle Soreness | Pre-Exercise (Day -1) to Post Exercise Recovery (up to 7 Days)
  100 mm visual analog scale from No Pain to Extreme Pain
Leg Strength Changes | Baseline to Day -1 Pre-Exercise (up to 4 Weeks)
  Change in Peak torque of maximum voluntary contraction (MVC)
Muscle Protein Synthesis | Post Exercise Day 1 to Day 7
  Change in Fractional Synthesis Rate
Muscle Protein Breakdown | Pre-Exercise (Day -1) to Post Exercise Recovery (up to 7 Days)
  Change in D3-3methylhistidine (D3-3MH)
Neuromuscular Function | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Change in Electromyography
Blood Biomarker Muscle Damage | Pre-Exercise (Day -1) to Post Exercise Recovery (up to 7 Days)
  Changes in blood biomarker of muscle damage
Blood Biomarker Oxidative Stress | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Changes in blood biomarker of oxidative stress

OTHER OUTCOMES:
Body Composition | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Changes in bioelectrical impedance analysis (BIA)
Muscle Biopsy Markers | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Change in muscle biopsy markers
Saliva Biomarkers | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Change in saliva biomarkers
Grip Strength | Baseline to Pre-Exercise Study Day -1 (up to 4 weeks)
  Change in hand grip dynamometer in kg
Microbiome | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Change in Alpha and Beta diversity
Short Physical Performance Battery (SPPB) Score | Baseline to Pre-Exercise Study Day -1 (up to 4 weeks)
  Change in 3 domains to assess functional mobility; Scores from 0 to 12 with higher scores indicating better mobility
Immunity Questionnaire | Baseline to Pre-Exercise Study Day -1 (up to 4 weeks)
  Participant reported information related to common cold symptoms
Quality of Life - Short Form 36 | Baseline to Pre-Exercise Study Day -1 (up to 4 weeks)
  Participant completed 36-item health survey resulting in a score from 0 to 100 where higher scores indicate better health status
Muscle Architecture | Baseline up to Post Exercise Study Day 7 (up to 5 weeks)
  Changes in ultrasound measurements

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Pereira, Study Chair — Abbott Nutrition
Locations (1):
- University of Nottingham, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No